CLINICAL TRIAL: NCT03810209
Title: Effect of Adding Magnesium Sulphate to Bupivacaine on the Quality of Ultrasound-guided Serratus Plane Block in Patients Undergoing a Modified Radical Mastectomy
Brief Title: SAP Block to Reduce Post Mastectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, clinical professor, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAP Block in Mastectomy
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2020-04

CONDITIONS: Serratus Anterior Plain Block
MeSH Terms: interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium sulphate group (Active Comparator): The investigator injected 28.5 mL of bupivacaine 0.5% and 1.5 ml MgSo4 (150 mg), a total volume of 30 ml, it was confirmed visually by the ultrasound.
  Interventions: Drug: Magnesium Sulphate
- control group (Placebo Comparator): The investigator injected 28.5 mL of Bupivacaine 0.5% and 1.5 mL of normal saline, a total volume of 30 ml, it was confirmed visually by the ultrasound.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Magnesium Sulphate — adding magnesium sulphate to local anaesthetic in SAP Block
  Other Names: MgSO4
  Arms: magnesium sulphate group
Drug: Normal saline — adding normal saline to local anaesthetic in SAP block
  Other Names: NaCl
  Arms: control group

SUMMARY:
To decrease post-operative pain in patients undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
The Serratus anterior Plane (SAP) Block has proven to be an effective component of multimodal analgesic regimens for a variety of thoracic procedures. It is designed to block primarily the thoracic intercostal nerves and to provide complete analgesia of the lateral part of the thorax and it may be a viable alternative to paravertebral blockade and thoracic epidural analgesia and may be associated with fewer side effects. It's straight forward to perform, with high success rate and minimal incidence of complications.

It was reported prolonged numbness over the area supplied by the lateral cutaneous branches of the T2-T9 spinal nerves using only 0.4 ml.kg-10.125% levobupivacaine. This is remarkable, because alternative techniques such as intercostal, interpleural and thoracic paravertebral block require relatively high concentrations and volumes of local anesthetics to produce similarly prolonged, multi-dermatomal thoracic analgesia.The duration of Serratus plane block is limited to the effect of administered local anesthetics (LAs). However, recently adjuvants such as epinephrine, ketamine and clonidine are added to LA solution in concentrations advocated for other peripheral blocks to prolong the effect of block with promising results.

Evidence supporting the presence of N-methyl-D-aspartate (NMDA) receptors in skin and muscles have led to the use of magnesium sulphate (MgSO4) (NMDA antagonist) via different routes for brachial plexus block and via neuraxial route. Until date, no study has been done to evaluate the role of MgSO4 as an adjuvant in SAP block. Therefore, the investigators intended this study to evaluate the role of MgSO4 as an adjuvant to bupivacaine in ultrasound (USG)-guided SAP block for postoperative analgesia in patients scheduled for modified radical mastectomy.

While the key requirement for successful regional anesthetic blocks is ensuring optimal distribution of local anesthetic around nerve structures, ultrasound guidance enables the anesthetist to secure an accurate needle position and to monitor the distribution of the local anesthetic in real time.

ELIGIBILITY:
Inclusion Criteria:

* Adult, female patients, ASA physical status I, II, and III aged older than 18 years scheduled for modified radical mastectomy surgery under general anesthesia.

Exclusion Criteria:

Any known allergies to the study drugs. Anatomical abnormalities or infections in the serratus region. Bleeding disorders e.g. thrombocytopenia, high INR, high PT in chronic liver or impaired kidney). Patients on chronic pain medications or regularly receiving analgesics. Pregnant or breast feeding patients. Body Mass Index (BMI) more than 35.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females with breast cancer for modified radical mastectomy
Enrollment: 40 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
The duration of analgesia measured by the time of first analgesic request | post operative 24 hours
  magnesium group showed delayed first analgesic request

CONTACTS AND LOCATIONS:
Overall Officials: abdelrhman alshawadfy, Principal Investigator — suez canal univesity
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No